CLINICAL TRIAL: NCT06675058
Title: Caries Location and Its Effect on the Success Rate of Indirect Pulp Treatment in Primary Molars: A Comparative Clinical Study
Brief Title: Caries Location and Its Effect on the Success Rate of Indirect Pulp Treatment in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yomna Hussein Moselhy Sayed Ahmed, Dr. Yomna Hussein Moselhy, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422023530604
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Deep Caries Lesion of Primary Teeth; Dental Pulp Diseases; Deep Proximal Caries; Deep Occlusal Caries; Reversible Pulpitis; Pulpitis; Decayed Teeth
Keywords: Indirect Pulp Treatment; IPT; Caries location; Caries Site; Proximal and occlusal Caries; Proximal Caries; Occlusal Caries; Pulp Therapy; Reversible Pulpitis; Pulpitis; deciduous teeth; Caries in milk teeth
MeSH Terms: conditions — Dental Pulp Diseases; Pulpitis; Dental Caries

STUDY DESIGN:
Intervention Model Description: a Selective Case Study ( Prospective Clinical Trial)
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary teeth with deep proximal caries (Experimental): In primary molars with deep proximal caries indirect pulp treatment will be performed by removing infected dentin while affected dentin in pulpal floor will be left in place. Teeth will be capped by a dressing material.
  Interventions: Procedure: Indirect Pulp Treatment
- Primary teeth with deep occlusal caries (Active Comparator): In primary molars with deep occlusal caries also IPT will be performed. Soft infected dentin will be carefully removed until the dried, hardened affected dentin with a leathery consistency reached then teeth will be capped by a dressing material
  Interventions: Procedure: Indirect Pulp Treatment

INTERVENTIONS:
Procedure: Indirect Pulp Treatment — Indirect pulp treatment is considered one of the most conservative pulp therapies, which preserves the pulp's vitality in teeth with reversible pulpitis. It has been chosen to be the intervention in both groups as the aim of this study is to assess the impact of caries location (proximal vs. occlusal caries) in influencing the success rate of IPT.

SUMMARY:
The following study will be created to evaluate how the location of caries affects the effectiveness of indirect pulp treatment in primary molars. aiding in the development of evidence-based recommendations for pediatric dentists.

DETAILED DESCRIPTION:
A selective case study design will be employed, focusing on primary molars with either occlusal or proximal carious lesions. Children aged between 3 to 7 years meeting the inclusion criteria will be examined clinically and radiographically to assess the extent and location of the carious lesion. Two groups will be involved in the study; primary molars will be submitted to each group based on whether the lesion is proximal or occlusal. Both groups will then receive indirect pulp therapy, and a clinical and radiographic evaluation for one year will be conducted.

The purpose of this study is to examine how the location of caries, whether proximal or occlusal, affects the success rate of IPT in primary molars. Understanding this relationship is essential for developing more tailored clinical approaches in pediatric dentistry to ensure long-term treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Participant criteria:

  1. Children aged between 3-7 years
  2. Children in complete physical and mental health.
  3. Children with free medical history.
  4. Patient with favorable attitudes, which will be assessed by using Frankl behavior rating.

Teeth criteria:

1. Primary molars with active occlusal or proximal deep caries.
2. Teeth with reversible pulpitis
3. Asymptomatic teeth or teeth with provoked pain of short duration
4. Teeth should be restorable.

Exclusion Criteria:

* Clinical signs or symptoms suggesting evidence of pulp degeneration or a non -vital tooth such as:

  * Clinical symptoms or history indicating irreversible pulpitis as (spontaneous pain, throbbing pain).
  * Tenderness to percussion.
  * Soft tissue swelling, abscess, draining fistula or sinus tracts.
  * Pathological Tooth mobility.

Presence of the following Radiographic criteria:

* Periapical or inter-radicular radiolucency.
* Internal or external pathological root resorption.
* Furcation involvement
* Widening of periodontal space.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate of primary molars with deep occlusal or proximal caries treated by Indirect Pulp Treatment (IPT) | one year follow up
  Clinical success rate will be assess through assessment of the following :
  Post-operative Pain (percentage of absence of pain), Presence or absence of clinical signs (e.g., swelling, abscess, sinus tract), and Pain on Percussion

SECONDARY OUTCOMES:
Radiographic success rate of primary molars with deep occlusal or proximal caries treated by Indirect Pulp Treatment (IPT). | one year follow up
  Radiographic Success Rate will be assess every (6, and 12 months) through assessment of the following in the x-ray film :
  No radiographic evidence of periapical or inter-radicular radiolucency, No internal or external root resorption, No furcation involvement, and No widening in the periodontal membrane ligament )

IPD SHARING:
Plan to Share IPD: Undecided